CLINICAL TRIAL: NCT03977233
Title: Impact of Tumor and Stromal Subtypes on Efficacy of Neoadjuvant FOLFIRINOX in Subjects With Non-Metastatic Pancreatic Cancer
Brief Title: Tumor Subtypes in Subjects on FOLFIRINOX With Non-Metastatic Pancreatic Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC1843
Record Dates: First submitted 2019-06-04; First posted 2019-06-06 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Pancreatic Ductal Adenocarcinoma (PDAC); Cancer of Pancreas; Pancreatic Cancer, Adult; Pancreas Adenocarcinoma; Pancreatic Neoplasms; Pancreatic Cancer Non-resectable; Pancreatic Cancer Resectable
Keywords: Pancreatic Ductal Adenocarcinoma; Pancreatic Cancer Non-resectable; Pancreatic Cancer Resectable; neoadjuvant FOLFIRNOX; FOLFIRINOX; Pancreatic Cancer, Adult
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatic cancer, adult | interventions — Oxaliplatin; Leucovorin; Irinotecan; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- SingleArm: FOLFIRINOX (Experimental): Subjects will receive FOLFIRINOX as an outpatient every 14 days per community standards of medical care. Protocol-based therapy will continue for 12 cycles (24 weeks) or until disease progression, unacceptable toxicity, study withdrawal, or subject death. Subjects will have the option of surgical resection after 8 cycles of therapy if repeat scans show evidence of resectable disease. The starting doses for mFOLFIRINOX regimen are: oxaliplatin 85 mg/m2, followed by leucovorin 400 mg/m2 given simultaneously with irinotecan 180mg/m2, followed by 5FU 400 mg/m2 bolus and then 2400 mg/m2 via continuous infusion.
  Interventions: Drug: Oxaliplatin; Drug: Leucovorin; Drug: Irinotecan Hydrochloride; Drug: 5-FU

INTERVENTIONS:
Drug: Oxaliplatin — 85 mg/m2 in 250 cc Dextrose solution given by IV on Day 1 of each 14-day cycle
  Other Names: Eloxatin
Drug: Leucovorin — 400 mg/m2 in 100 cc dextrose solution given with irinotecan by IV on Day 1 of each 14-day cycle
  Other Names: folinic acid
Drug: Irinotecan Hydrochloride — 180 mg/m2 in 500cc dextrose solution given with leucovorin by IV on Day 1 of each 14-day cycle
  Other Names: Camptosar
Drug: 5-FU — 400 mg/m2 bolus and then 2400 mg/m2 via continuous infusion on Day 1 of each 14-day cycle
  Other Names: Adrucil

SUMMARY:
This is a research study to evaluate how the genetic makeup of Pancreatic Ductal Adenocarcinoma (PDAC) can affect the response to FDA-approved chemotherapy treatment, FOLFIRINOX, given before surgery to remove the tumor. Certain types of PDAC tumors can be surgically resected (removed). However, not all types of PDACs are resectable, especially if they are close to important structures like blood vessels or intestines. These types of PDACs are treated with chemotherapy such as FOLFIRINOX. Research studies showed that chemotherapy after surgical resection of PDAC tumors reduced the risk of the cancer returning.

Chemotherapy is used to treat PDAC that has not spread outside of the pancreas and is not resectable. FOLFIRINOX is a chemotherapy treatment that combines multiple chemotherapeutic agents, including oxaliplatin, leucovorin, irinotecan, and 5-FU. Patients receive these agents by intravenous infusion. Of these drugs, 5-FU requires you to return home with a chemotherapy pump that will deliver chemotherapy over 46 hours. This regimen has been studied in pancreatic cancer that has been removed with surgery as a method for preventing the cancer from returning. Studies showed FOLFIRINOX chemotherapy reduced the risk of cancer returning and increased patients survival. In this study, researchers want to know if FOLFIRINOX chemotherapy given before surgery will make the cancer easier to remove with surgery and increase the chances of the cancer staying away after surgery.

Researchers have shown that pancreatic cancers are not all the same when you look at the DNA and RNA that is inside a pancreatic cancer cell.

Depending on the expression of different genes in a cancer cell, some pancreatic cancers may respond differently to chemotherapy. In this study researchers want to know if FOLFIRINOX chemotherapy can change the genetic profile of the cancer. This will be studied by obtaining a biopsy of the cancer before the start of chemotherapy, and after 8 treatments of chemotherapy. They will also study cancer cells that will be collected from blood samples.

DETAILED DESCRIPTION:
This is a single arm, phase II clinical trial designed to assess the impact of tumor and stromal molecular subtypes on the efficacy of neoadjuvant FOLFIRNOX in untreated subjects with resectable, borderline resectable and unresectable locally advanced pancreatic ductal adenocarcinoma (PDAC). Subjects will undergo an EUS-guided core biopsy of the pancreas prior to treatment and after cycle 8 of FOLFIRINOX. Imaging will be performed after every 4 cycles of chemotherapy (8 weeks) and reassessed for resectability after 12 cycles. If patients show a response to treatment that is deemed by the surgical oncologist to be amenable to resection, surgery can be pursued after 8 cycles of therapy. In this case, the remaining 4 cycles of treatment will be given after surgery.

Duration of Therapy:

In the absence of treatment delays due to adverse events, treatment may continue until:

* Disease progression,
* Inter-current illness that prevents further administration of treatment,
* Unacceptable adverse event(s),
* Subject decides to withdraw from the study, or
* General or specific changes in the subject's condition render the subject unacceptable for further treatment in the judgment of the investigator.

Duration of Follow Up:

- Subjects will be followed for 36 months after removal from study treatment or until death, whichever occurs first. Subjects removed from study treatment for unacceptable adverse events will be followed until resolution or stabilization of the adverse event.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained to participate in the study and HIPAA authorization for release of personal health information.
* Histologically or cytologically confirmed adenocarcinoma of the pancreas with no evidence of distant metastatic disease.
* Subject has no evidence of co-morbidities precluding the potential to undergo surgical resection of PDAC as determined by surgical investigator.
* Subjects must be willing to undergo a mandatory pre- and post-treatment EUS guided core biopsy of the pancreatic mass.
* Measurable or non-measurable but evaluable (as determined by Response Evaluation Criteria in Solid Tumors version 1.1 [RECIST 1.1]) resectable, borderline resectable or unresectable locally advanced PDAC.
* Subject has adequate performance status as defined by ECOG performance status 0 or 1.
* Subject has received no prior chemotherapy or chemoradiotherapy for pancreatic cancer. Subjects have not previously received surgery to remove pancreatic cancer.
* Age ≥ 18 years of age.
* Subject has adequate organ function at study entry.
* Subject has life expectancy of at least 6 months.

Exclusion Criteria:

* Subject has any evidence of local recurrence or metastatic pancreatic cancer.
* Other malignancies within the past 5 years except for adequately treated cervical or vulvar carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors (Ta, Tis and T1).
* Subject has hypersensitivity to 5FU, oxaliplatin or other platinum agent, or irinotecan or to their excipients.
* Subject has known dihydropyrimidine dehydrogenase (DPD) enzyme deficiency.
* Participation in any investigational drug study within 4 weeks preceding the start of study treatment. Subjects are not permitted to participate in another investigational drug study while being treated on this protocol. Subjects participating in other clinical trials that are receiving SOC FOLFIRINOX are permitted on study.
* Subject has current evidence of any condition that makes participating in this study not in the best interest of the subject, including but not limited to:

  * Myocardial infarction within the past 6 months
  * New York Heart Association (NYHA) Class III or IV heart disease
  * Active infection requiring IV antibiotics
* Subject has a history of or suspected Gilbert's syndrome or known homozygosity for UGT1A1*28 polymorphism (baseline testing not required).
* Subject has sensory peripheral neuropathy grade ≥ 2.
* Major surgery, open biopsy or significant traumatic injury within 4 weeks of first study drug.
* Subject is unable or unwilling to discontinue use of ketoconazole or St John's wort. Use of phenytoin, carbamazepine, phenobarbital, rifampin and rifabutin is discouraged, but not contraindicated. If subjects require phenytoin, carbamazepine or phenobarbital monitoring of drug levels is suggested during the study.
* Subject is pregnant or lactating.
* Psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the subject before registration in the trial.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2019-06-12 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Best disease control rate by Pancreatic ductal adenocarcinoma (PDAC) subtype | 6 months after start of treatment
  To evaluate the association between PDAC tumor subtype (particularly basal-like versus classical subtype) and best disease control rate (DCR) after administration of FOLFIRINOX in subjects with non-metastatic pancreatic cancer, DCR is defined as the proportion of patients with either Complete Response (CR), partial response (PR), or stable disease (SD) as determined by RECIST 1.1, Response Evaluation Criteria In Solid Tumors Criteria. CR is defined as disappearance of all target lesions; PR as a >=30% decrease in the sum of the longest diameter of target lesions; and SD as no response or less response than Partial or Progressive.

SECONDARY OUTCOMES:
Rate of resectability | 6 months after the start of treatment
  The number of patients who following treatment with FOLFIRINOX were subsequently deemed to have resectable disease and underwent surgical resection
Overall survival | 3 years
  median overall survival (OS) of all patients receiving FOLFIRINOX on study as well as in 1) resectable, 2) borderline resectable and 3) unresectable PDAC, measured from the start of treatment until death from any cause.
Progression free survival | 3 years
  Median time from start of treatment until death or progression as defined by RECIST 1.1 Criteria, for all patients and with respect to each tumor and stroma subtype. Progressive Disease (PD), is defined as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
best objective response rate (ORR; complete response (CR) + partial response (PR)) | 6 months from start of study treatment
  Estimation of the best ORR for all patients and with respect to each tumor and stroma subtype. ORR is defined as the proportion of patients with either Complete Response (CR) or partial response (PR) as determined by RECIST 1.1, Response Evaluation Criteria In Solid Tumors Criteria. CR is defined as disappearance of all target lesions; PR as a >=30% decrease in the sum of the longest diameter of target lesions;
rate of drug-related grade 3 to 5 adverse events | 6 months from the start of treatment
  rate of drug-related grade 3 to 5 adverse events, assessed based upon patient reported toxicity as measured by the NCI Common Terminology Criteria for Adverse Events (CTCAE v5.0). The CTCAE is a descriptive terminology which can be utilized for Adverse Event (AE) reporting. A grading (severity) scale is provided for each AE term. Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental Activities of Daily Living (ADL). Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL. Grade 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to AE.
R0 resection rate | 6 months from start of treatment
  The number of patients who underwent surgical resection and whose surgical specimens had a microscopically margin-negative resection (R0).
proportion of patients whose tumor/stroma subtype changes after treatment with FOLFIRINOX | 6 months from start of treatment
  The proportion of patients whose tumor/stroma subtype changed from baseline after treatment with FOLFIRINOX. This will be calculated separately for tumor and stroma.

CONTACTS AND LOCATIONS:
Overall Officials: Ashwin Somasundaram, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials